CLINICAL TRIAL: NCT05249803
Title: "Clinical Characteristics, Comorbidities and Outcome of Critically Sick Patients With COVID-19 Pneumonia Admitted in Intensive Care Unit of a Tertiary Care Hospital in Lahore, Pakistan": A Retrospective Cohort Study
Brief Title: "Clinical Characteristics, Comorbidities and Outcome of Critically Sick Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: FMH College of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Aijaz Zeeshan Khan Chachar, Consultant Physician (Senior Registrar), FMH College of Medicine and Dentistry
Other Study IDs: FMH-27/12/2021-IRB-983
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia
Keywords: Comorbidities; Outcomes; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with COVID-19 pneumonia: These patients were admitted in ICU for management of Covid-19 pneumonia usual care was offered to all patients
  Interventions: Combination Product: Patients with COVID-19 Pneumonia

INTERVENTIONS:
Combination Product: Patients with COVID-19 Pneumonia — Patients were offered with usual care of COVID-19 in ICU and we did retrospective study

SUMMARY:
COVID-19, caused by severe acute respiratory syndrome corona virus 2 (SARS-CoV-2), is a multisystem disease which primarily involves the respiratory tract. The first case of COVID-19 was identified in late 2019 in the province of Wuhan, China which was followed by the rapid spread of the disease globally, becoming a present-day pandemic.

Objectives: The aim of this study was to describe the clinical characteristics, comorbidities and outcome of the critically sick patients with COVID-19 pneumonia admitted in ICU of a tertiary care hospital in Lahore.

DETAILED DESCRIPTION:
Objectives: The aim of this study was to describe the clinical characteristics, comorbidities and outcome of the critically sick patients with COVID-19 pneumonia admitted in ICU of a tertiary care hospital in Lahore.

Material & Methods:

Study design: Retrospective study. Study Settings: Study was conducted in Fatima Memorial Hospital, Lahore. Study Duration: Study was conducted on Covid-19 patients who were admitted from March 2021 to August 2021.

ELIGIBILITY:
Inclusion Criteria:

* Critically sick patients with COVID-19 Pneumonia
* All admitted ICU patients with a diagnosis of COVID-19 pneumonia
* Patients having positive reverse transcriptase PCR for COVID-19
* Patients with High-resolution computed tomography (HRCT) chest findings suggestive of COVID-related lung injury
* All patients above 16 years of age with both genders( males and females)

Exclusion Criteria:

* All patients with PCR negative with mild symptoms
* Patients with No signs of COVID-19 pneumonia on HRCT chest

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-interventional retrospective cohort study of critically sick patients with COVID-19 pneumonia admitted in the Intensive Care Unit of Fatima Memorial hospital (FMH) in Lahore, Pakistan from March 2021 to August 2021 4.3. Sample Size & Technique: Records of 133 patients admitted to the ICU of the Fatima memorial hospital, Lahore, were studied.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  The primary endpoint of the study will be to assess the ICU mortality (in percentages% and Numbers) of critically sick patients with COVID-19 pneumonia admitted to the intensive care unit

SECONDARY OUTCOMES:
Comorbidities | 6 months
  we will assess various comorbidities in critically sick patients with COVID-19 pneumonia admitted to the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Aijaz Zeeshan K Chachar, MBBS,FCPS, Principal Investigator — FMH College of Medicine & Dentistry
Locations (1):
- Fatima Memorial Hospital College of Medicine & Dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All the record can be retrieved from medical record department of fatima memorial hospital Lahore
Supporting Information: Study Protocol, SAP, ICF
URL: http://www.fatimamemorial.org.pk